CLINICAL TRIAL: NCT03856645
Title: A Phase 2, Multi-centeR, Randomized, DoUBle-Masked, Placebo-Controlled StudY to Evaluate the Clinical Safety and Efficacy of OKG-0301 in the Treatment of Acute Adenoviral Conjunctivitis
Brief Title: OKG-0301 for the Treatment of Acute Adenoviral Conjunctivitis
Acronym: RUBY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Okogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OKO-210
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- OKG-0301 0.012% w/v (Experimental)
  Interventions: Drug: OKG-0301
- OKG-0301 0.03% w/v (Experimental)
  Interventions: Drug: OKG-0301
- Vehicle Control (Placebo Comparator)
  Interventions: Drug: OKG-0301

INTERVENTIONS:
Drug: OKG-0301 — OKG-0301 is an experimental ophthalmic antiviral and immunomodulatory therapeutic

SUMMARY:
Acute adenoviral conjunctivitis is a highly contagious, widespread endemic disease associated with frequent outbreaks, significant patient discomfort, lost productivity, and in some cases permanent visual compromise from long-term immune mediated sequelae. OKG-0301 is a novel ophthalmic solution with a potent ribonuclease that has broad-spectrum antiviral properties relevant for the treatment of acute adenoviral conjunctivitis. This randomized, double masked, multi-center Phase 2 study is being conducted entirely within Australia and is designed to support the safety and efficacy of OKG-0301 for the treatment of acute adenoviral conjunctivitis. The study intends to show superiority of OKG-0301 Ophthalmic Solution compared to vehicle for the primary efficacy endpoint of mean change from baseline in viral titre in patients with acute adenoviral conjunctivitis. Secondary efficacy endpoints including adenoviral eradication, clinical cure of acute adenoviral conjunctivitis, subepithelial infiltrates, other clinical signs and symptoms, and rate of cross-over infection to the other eye will also be assessed. Safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Each patient MUST:

1. Be willing and able to provide informed consent either written, or if the patient is not able to read, provide consent as stipulated by local laws and Human Research Ethics Committee (HREC) guidelines.
2. Be willing and able to follow all instructions and attend all study visits.
3. Have a clinical diagnosis of suspected acute adenoviral conjunctivitis in at least 1 eye and the presence of both of the following minimal clinical signs in that same eye:

   * Bulbar conjunctival redness: a minimum grade of '1' on 0-3 scale
   * Watery ocular discharge: a minimum grade of '1' on a 0-3 scale
4. Patient reported presence of signs and symptoms consistent with adenoviral conjunctivitis equal to or less than 3 days in same eye prior to Visit 1.
5. Have a positive AdenoPlus® test at Visit 1 in the same eye that meets the minimum 1+ grade for bulbar conjunctival redness and watery ocular discharge.
6. Be willing to discontinue contact lens wear for the duration of the study.

Exclusion Criteria:

Each patient MUST NOT:

1. Have known sensitivity or poor tolerance to any component of the study medications or diagnostics.
2. Have a history of ocular surgical intervention or trauma within 12 weeks prior to Visit 1 or planned for the period of the study.
3. Have presence of any active ocular inflammation (e.g., uveitis, allergic conjunctivitis, ocular rosacea, or iritis), other than acute adenoviral conjunctivitis.
4. Have clinical signs or presence of an ocular infection other than acute adenoviral conjunctivitis (e.g., bacterial, fungal or other ocular viral infection, such as herpes).
5. Have the presence of corneal subepithelial infiltrates at baseline.
6. Have a history of recurrent corneal erosion syndrome, ulcerative keratitis or dry eye, including meibomian gland dysfunction and other ocular surface diseases.
7. Have presence of blepharitis, lid abnormality, significant inflammation of the lid margin, or ptosis.
8. Have lacrimal duct obstruction in either eye.
9. Have presence of any other clinically significant findings during the slit lamp exam that may interfere with study parameters or otherwise confound the data as determined by the investigator
10. Have any clinically significant retinal or optic nerve findings (as observed in the non-dilated fundus exam) or prior diagnoses in either eye that may interfere with study parameters or otherwise confound the data as determined by the investigator).
11. Have used any topical ocular or systemic anti-viral or topical ocular or systemic corticosteroid within 7 days of enrollment and do not plan to start any topical ocular or systemic anti-viral during study duration. Inhaled, intranasal, and topical dermatologic steroids (except on the face) are allowed during the study.
12. Initiate or continue the use of warm or cold compresses for the duration of the trial.
13. Have used any topical ophthalmic solutions, including tear substitutes and diagnostics, within 2 hours of Visit 1 and be unable to discontinue all topical ophthalmic solutions (including diagnostics, except as required by this protocol and antibiotics) for the duration of the study. In addition, if the patient has used an artificial tear or other topical ophthalmic formulated in a hydrogel within the past 72 hours.
14. Be currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive pregnancy test.
15. Have any uncontrolled (not on a stable regimen for the past 30 days) systemic disease or debilitating disease (e.g., cardiovascular disease, hypertension, diabetes, or cystic fibrosis) or taking medications known to impact the ocular surface and/or tear film.
16. Have a planned overnight hospitalization during the period of the study.
17. Have any uncontrolled (not on a stable regimen for the past 30 days) autoimmune disease or taking medications known to impact the ocular surface and/or tear film.
18. Have prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device.
19. Have a condition or a situation which, in the investigator's opinion, may put the patient at increased risk, confound study data, or interfere significantly with the patient's study participation.
20. Be unlikely to follow study instructions or to complete all required study visits or has a condition or situation that in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in viral titre levels in the study eye | Day 7
  PFU

SECONDARY OUTCOMES:
Clinical Cure as Measured by the Absence of Bulbar Conjunctival Injection | Day 4, 7 and 14
  Clinical cure of acute adenoviral conjunctivitis as measured by the absence (score = 0) of bulbar conjunctival redness (graded using the validated Ora Calibra Scale 16.2: Bulbar Conjunctival Redness Grading Scale)
Clinical Cure as Measured by the Absence of Watery Conjunctival Discharge | Day 4, 7 and 14
  Clinical cure of acute adenoviral conjunctivitis as measured by the absence (score = 0) of watery conjunctival discharge (graded on a scale of 0-3 based on severity, developed specifically for this trial)
Adenoviral eradication (CC-IFA) | Day 4, 7 and 14
  Adenoviral eradication is defined as negative CC-IFA. CC-IFA will be conducted using conjunctival swab samples collected at each visit to determine the presence or absence of adenovirus.
Adenoviral eradication (PFU) | Day 4, 7 and 14
  Adenoviral eradication is defined as zero plaques in cultures of ocular samples. PFU will be conducted using conjunctival swab samples collected at each visit to determine the presence or absence of adenovirus.
Severity of subepithelial infiltrates | Day 4, 7 and 14
  Evaluation of SEIs in study eye, assessed under slit lamp exam with Investigator grading on a 0-3 semi-quantitative scale (developed specifically for this study).
The rate of cross-over infection | Day 4, 7 and 14
  Clinical signs in contra-lateral eye that initially presented with no signs or symptoms of adenoviral conjunctivitis

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Albury Eye Clinic, Albury, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - The Royal Adelaide Hospital, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
  - The Royal Victorian Eye and Ear Hospital, Melbourne E., Victoria
  - Lions Eye Institute Day Surgery Centre, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No